CLINICAL TRIAL: NCT03571074
Title: Hyperoxia Before and After Cardiac Arrest and Myocardial Damage, a Retrospective Cohort Study
Brief Title: Hyperoxia Before and After Cardiac Arrest and Myocardial Damage
Status: Completed | Type: Observational
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Kathrine Schmidt Groenbek, Research Assistant, Bispebjerg Hospital., University Hospital Bispebjerg and Frederiksberg
Other Study IDs: HyperoxiaandCardiacarrest
Record Dates: First submitted 2018-06-04; First posted 2018-06-27 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hypoxia: Defined as a group of patients with oxygen saturation <94 % irrespective of supplemental oxygen.
  If COPD, defined as oxygen saturation <88 % irrespective of supplemental oxygen.
  Interventions: Other: Oxygenation
- Normoxia: Defined as a group of patients with oxygen saturation 94 % - 98 % in combination of supplemental oxygen, or oxygen saturation >94 % without supplemental oxygen.
  If COPD, defined as oxygen saturation 88 % - 92 % in combination of supplemental oxygen, or oxygen saturation >88 % without supplemental oxygen.
  Interventions: Other: Oxygenation
- Hyperoxia: Defined as a group of patients with oxygen saturation >98 % in combination of supplemental oxygen.
  If COPD, defined as oxygen saturation >92 % in combination of supplemental oxygen.
  Interventions: Other: Oxygenation

INTERVENTIONS:
Other: Oxygenation — Oxygenation measured as oxygen supply and saturation before cardiac arrest, and oxygenation measured as PaO2 after cardiac arrest.

SUMMARY:
Several studies show how patients with hyperoxia after cardiac arrest has increased mortality, but the association of hyperoxia before cardiac arrest and myocardial damage has never been investigated. Neither has the association between hyperoxia after cardiac arrest and myocardial injury.

Our research hypothesis is that hyperoxia before cardiac arrest aggravates myocardial damage, secondly we wish to analyze the association between hyperoxia after cardiac arrest and myocardial injury.

The exposure variables is oxygenation within 48 hours before and 48 hours after cardiac arrest, our primary outcome is myocardial damage and will be measured as peak troponin within 30 days after cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* With a record of ICD-10 diagnosis of cardiac arrest in 2014, admitted to a hospital in the Capital Region of Denmark.
* First recorded cardiac arrest in 2014
* Admitted to ICU
* Serum troponin measured within 7 days after cardiac arrest

Exclusion Criteria:

* Out of hospital cardiac arrest, OHCA
* In of hospital cardiac arrest, IHCA, but with no registered saturation before cardiac arrest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with in hospital cardiac arrest, who had return of spontaneus circulaiton and was then admitted to ICU in a hospital in the Capital Region of Denmark.
Sampling Method: Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Peak troponin within 30 days after cardiac arrest | 30 days
  Troponin measurements on patients after cardiac arrest.

SECONDARY OUTCOMES:
30-day and 1-year mortality | Up to 1 year.
Troponin area under the curve within 3 days after cardiac arrest | 3 days
Length of ICU stay after cardiac arrest | through study completion,on average of 4-8 weeks.
Length of hospital stay after cardiac arrest | through study completion,on average of 4-8 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided